CLINICAL TRIAL: NCT06612294
Title: A Randomized Trial of Perception of Airflow Limitation Training to Improve Outcomes for Older Adults With Asthma
Brief Title: Asthma Symptom Perception Study
Acronym: ASP RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Albert Einstein College of Medicine (Other); Yeshiva University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Juan Wisnivesky, Division Chief, General Internal Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 23-0259; 1R01HL171676-01 (NIH)
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Research Coordinators conducting interviews and all investigators will be blinded to treatment allocation. Project staff will be assigned as Care Coaches for the intervention and the control treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PEF group with active booster (Experimental): This arm will have 3 intervention sessions over 6 weeks and an additional (active) session at 6-month time point.
  Interventions: Behavioral: PEF Interventional Session; Behavioral: Active booster
- PEF group with control booster (Experimental): This arm will have 3 intervention sessions over 6 weeks and a control booster session at the 6-month time point.
  Interventions: Behavioral: PEF Interventional Session; Behavioral: Control Booster
- Control Group (Placebo Comparator): This arm will have 3 control sessions over 6 weeks and a control booster session at 6-month time point.
  Interventions: Behavioral: Control Sessions; Behavioral: Control Booster

INTERVENTIONS:
Behavioral: PEF Interventional Session — 3 sessions over 6 weeks for asthma management
  Arms: PEF group with active booster; PEF group with control booster
Behavioral: Control Sessions — 3 sessions over 6 weeks for asthma management
  Arms: Control Group
Behavioral: Control Booster — A single booster session after the 6-months assessments are completed.
  Arms: Control Group; PEF group with control booster
Behavioral: Active booster — A single booster session after the 6-months assessments are completed.
  Arms: PEF group with active booster

SUMMARY:
Asthma affects 8% of the United States population ages >60 years and causes considerable harm: older adults are 4 times more likely to die from asthma and have twice the risk of hospitalization. The burden of asthma is notably greater among minoritized older adults. Research suggests that perception of expiratory airflow limitation may be a major determinant of asthma outcomes in older adults, and that older adults are substantially less aware of airway obstruction than younger adults. These observations suggest that perception of airflow limitation is a potential target for improving outcomes of older patients with asthma. The research team completed a pilot randomized controlled trial (RCT) of an intervention that trains older adults with asthma to better perceive expiratory airway obstruction through feedback via peak expiratory flow (PEF) prediction and couples this feedback with motivational interviewing (MI) to promote change in asthma self-management behaviors. Compared to an attention control, the intervention improved PEF, perception of airflow limitation and asthma control. In this project, the research team will conduct a fully powered RCT to test the intervention's efficacy among 300 adults ages ≥60 years with uncontrolled asthma who are on controller medications (daily maintenance or as needed) recruited from underserved inner-city medical practices in New York City. Patients will be randomized to the intervention or a time and attention matched educational control. The intervention and control will be delivered in 3 sessions over 6 weeks. The study will test the impact of the intervention on perception of expiratory airflow limitation in older adults with asthma, examine the efficacy of the intervention for improvements in lung function (PEF), self-reported asthma control (Asthma Control Questionnaire [ACQ] scores), quality of life (Asthma Quality of Life Questionnaire [AQLQ] scores), and emergency department and hospital use, and test the intervention's impact on mean daily ICS dose used (daily maintenance and as needed). Data will be collected at baseline, 1-month, 6-months (primary analyses of effectiveness) and 12-months post-intervention. In secondary analyses, the research team will test the sustainability of treatment effects with vs. without the booster treatment session (active booster vs. attention control booster) delivered immediately after the 6-month assessment on outcomes at 12-months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* English or Spanish speaking
* Self-report or physician diagnosis of asthma >1 year ago
* Uncontrolled asthma

Exclusion Criteria:

* Dementia
* Chronic obstructive pulmonary disease (COPD), or other chronic respiratory illnesses,
* Congestive Heart Failure (CHF, New York Heart Association [NYHA] stages 4-5)
* Cigarette smoking >15 packs-years

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2028-12-22 (Estimated); Study Completion 2028-12-22 (Estimated)

PRIMARY OUTCOMES:
Peak expiratory flow (PEF) Values | at baseline, 1-month, 6-months, and 12-months post-intervention
  Perception accuracy of airflow limitation will be measured by perceived and actual PEF values.
Mean daily ICS dose used | at baseline, 1-month, 6-months, and 12-months post-intervention
  Mean daily ICS dose will be recorded for asthma medications

SECONDARY OUTCOMES:
Number of participants using medications on ≥70% of days prescribed | at baseline, 1-month, 6-months, and 12-months post-intervention
  Adherence will be measured via the number of participants using medications on ≥70% of days prescribed.
Participant personal best PEF percent | at baseline, 1-month, 6-months, and 12-months post-intervention
  Participant personal best PEF percent will be collected using the AM2 during assessments of perception of airflow limitation.
Asthma Control Questionnaire [ACQ] scores | at baseline, 1-month, 6-months, and 12-months post-intervention
  The ACQ is a self-reported questionnaire that assess asthma beliefs about asthma control. The ACQ is an instrument, full scale from 0-6, higher score indicates more impairment.
Asthma Quality of Life Questionnaire [AQLQ] scores | at baseline, 1-month, 6-months, and 12-months post-intervention
  The AQLQ assess asthma beliefs about asthma quality of life. The AQLQ is an instrument, full scale from 1-7, higher score indicates better health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Wisnivesky, MD, DrPH, Principal Investigator — Division Chief, General Internal Medicine
Locations (2):
- United States (2):
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The research team will provide data sets and associated documents to the NIH study Program Official within timelines described in the NIH Policy for Data Sharing from Clinical Trials and Epidemiological Studies - no later than 3 years after the end of the clinical activity (final patient follow-up, etc.) or 2 years after the main paper of the clinical trial has been published - whichever comes first.
Access Criteria: Anyone who wishes to access the data. The research team will prepare public use, de-identified datasets which will be uploaded to the Inter-university Consortium for Political and Social Research (ICPSR) repository once the main study aims manuscripts have been published.